CLINICAL TRIAL: NCT02561897
Title: Efficacy and Safety of Edoxaban or Warfarin Therapy In Cardiovascular Implantable Electrical Device Procedures in Patients With Non-valvular Atrial Fibrillation
Brief Title: EdoxabaN or Warfarin Therapy In Device Procedures in Patients With Non-Valvular Atrial Fibrillation
Acronym: ENTICED-AF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not meet enrolment target for phase 1
Sponsor: Electrophysiology Research Foundation (Other)
Collaborators: Axio Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPRF2015-01
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental): Edoxaban 30 or 60 mg
  Interventions: Drug: Edoxaban
- Warfarin (Active Comparator): Warfarin 1 -1 0 mg
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Edoxaban
  Other Names: Savaysa
  Arms: Edoxaban
Drug: Warfarin
  Arms: Warfarin

SUMMARY:
This is a prospective randomized comparative evaluation of Edoxaban and Warfarin for safety and efficacy in perioperative use in patients with non-valvular atrial fibrillation (AF) undergoing clinically indicated implantation or replacement of cardiovascular implantable electrical devices.The primary objective is to compare the rates of local and systemic bleeding in subjects randomized to Edoxaban compared to subjects randomized to continuous warfarin in within 30 days of cardiac rhythm device implant with concomitant non-valvular AF.

DETAILED DESCRIPTION:
This is a prospective randomized comparative evaluation of Edoxaban and Warfarin for safety and efficacy in perioperative use in patients with non-valvular atrial fibrillation undergoing clinically indicated implantation or replacement of cardiovascular implantable electrical devices. This study is a randomized, open label, active-controlled trial with an open-label safety extension, designed to compare local and systemic bleeding within 30 days of cardiac rhythm device implant among subjects randomized to continuous Warfarin or interrupted (<24 hours) Edoxaban. The study will have three phases, a run in phase to establish stable warfarin therapy, an acute open label 30 day phase when subjects will be randomized in a 1:1 ratio to receive interrupted edoxaban or continuous warfarin followed by an open label follow up phase for an additional 5 months for safety monitoring. Drug transitions will be performed according to approved drug labeling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with established atrial fibrillation (AF) and bradycardia on long term (>3 weeks) therapeutic oral anticoagulant (OAC) with warfarin or another OAC who are undergoing new pacemaker system implant or existing pacemaker system revision.
* Subjects with newly detected bradycardia -tachycardia syndrome and AF who have been recently (less than 3 weeks) started on warfarin, have a therapeutic international normalized ratio (INR) and no thrombus on trans-esophageal echocardiogram (TEE) who are undergoing a new pacemaker system implant or revision.
* Subjects with AF and ventricular tachyarrhythmias (VT or VF) or acquired structural heart disease who are candidates for implantable cardioverter-defibrillator (ICD) therapy and are on long term (>3 weeks) therapeutic OAC with warfarin or another OAC who are undergoing new ICD system implant or existing ICD system revision.
* Subjects with newly detected AF with VT or VF who have been recently (less than 3 weeks) started on warfarin, have a therapeutic INR and no thrombus on TEE who are undergoing ICD system implant or revision

Exclusion Criteria:

* Clinically significant valvular heart disease
* Subjects requiring cardiovascular implantable electrical device (CIED) lead extraction e.g. for device site infection, endocarditis, leads under advisory or other conditions warranting lead(s) system extraction.
* Recent (<1 month) myocardial infarction
* Documented left atrial (LA) thrombus on TEE
* Contraindications to anticoagulant therapy or adverse event with prior warfarin or edoxaban therapy
* Creatinine clearance <30ml/min or >95 ml/min
* Hepatic disease, advanced
* Recent stroke (<3 months) or thromboembolic event
* Recent (<3months) intracranial or other major bleeding event
* Use of concomitant dual antiplatelet therapy or other oral, subcutaneous or parenteral anticoagulant therapy
* Subjects on warfarin without therapeutic INR levels before study entry
* Subjects with other clinically significant medical condition
* Subjects with life expectancy < 1 year
* Lead extraction procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Saksena, MBBS MD, Study Chair — Electrophysiology Research Foundation
Locations (1):
- Electrophysiology Research Foundation, Warren Township, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 2015-2017
  Recruited in hospital and medical clinic
Groups:
- Edoxaban: Edoxaban 30 or 60 mg
  Edoxaban
- Warfarin: Warfarin 1 -1 0 mg
  Warfarin
Period: Overall Study
Arm/Group | Edoxaban | Warfarin
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Warfarin | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.4) | 72.0 (12.5) | 69.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding
Description: Major local or systemic bleeding as defined in the protocol at 30 days after implant procedure
Time Frame: Within 30 days of procedure
Measure: Count of Participants; unit: Participants
Groups:
- Warfarin: One patient had a hematoma
- Edoxaban: No patient met primary outcome
Arm/Group | Warfarin | Edoxaban
Number analyzed (Participants) | 3 | 2
Participants | 1 | 0

2. Secondary Outcome: Thromboembolic and Cardiovascular Events
Description: Thrombotic events (embolism or stroke) through 6 months following the procedure in the Edoxaban and Warfarin groups and the rates of MACE events through 6 months following the procedure in the Edoxaban and Warfarin groups
Time Frame: Within 6 months of procedure
Measure: Count of Participants; unit: Participants
Groups:
- Warfarin; Edoxaban: No patient had secondary outcome
Arm/Group | Warfarin | Edoxaban
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Warfarin: To maintain therapeutic INR level
- Edoxaban: 60 mg tablet once daily
Arm/Group | Warfarin | Edoxaban
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin (N=3) | Edoxaban (N=2)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Superficial wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Superficial skin infection at three month follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02561897/Prot_SAP_000.pdf